CLINICAL TRIAL: NCT01428999
Title: Effects of Probiotics on Improving the Gastrointestinal Function and Intestinal Bacterial Flora
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BR-100-039
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-06

CONDITIONS: Gastrointestinal Function; Intestinal Bacteria Flora
Keywords: probiotics; gastrointestinal function; intestinal bacteria flora
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotics (Experimental): 1 pack bid use for 3 weeks
  Interventions: Dietary Supplement: probiotics
- Placebo (Placebo Comparator): placebo 1pack bid for 3 weeks
  Interventions: Dietary Supplement: probiotics

INTERVENTIONS:
Dietary Supplement: probiotics — probiotics 1 pack (2g) bid for three weeks

SUMMARY:
The purpose of this study is to evaluate the effect of "combined probiotics" to improve the gastrointestinal function and intestinal bacteria flora

DETAILED DESCRIPTION:
Probiotics were known to improve gastrointestinal function before. This is a single-blind placebo control clinical study. We will perform gastrointestinal function questionnaire and collect stool as baseline data before the study (0-week). Then healthy subjects will be randomized to two groups.

Experimental: probiotics 1 pack bid for 3 weeks. Probiotics : (AB-kefir)：Lactobacillus acidophilus,Bifidobacterium longum,Lactobacillus paracasei,Lactobacillus rhamnosus,Lactobacillus fermentum,Streptococcus thermophilus,Lactobacillus helveticus,Kluyveromyces fragilis. Other components include starch,oligosaccharide,yeast powder, superior standard spice， calcium pantothenate， VitB1， VitB12， biotin and folic acid.

Placebo group: placebo 1 pack bid for 3 weeks. Placebo: Except the probiotics (AB-kefir),the other components are the same with study group.

Then gastrointestinal function questionnaire and stool collection will be performed at the end of 1st, 2nd, 3rd, and 4th weeks after starting the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people who are aged between 20 and 40 years

Exclusion Criteria:

* 1. People who use probiotics medication and food that can inhibit bacteria growth within one month before the study 2. People who have active infection 3. People who have active or chronic gastro-intestinal disease 4. People who have diarrhea within two weeks before the study 5. People who are drug or alcohol abuser 6. People who are poor compliance

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Changes of gastrointestinal function after probiotics use | 28 days
  Changes of gastrointestinal function, such as constipation, abdominal distension and appetite after proiotics and placebo use.

SECONDARY OUTCOMES:
Changes of intestinal bacteria flora after probiotics use | 28 days
  1. Changes of intestinal bacteria flora: (1) aerobic bacteria count (2) anaerobic bacteria count (3) Bifidobacterium count (4) Clostridium perfringens count (5) Staphylococcus aureus count (6) E. coli and K. pneumoniae count
  2. The ratio for the antibiotics resistant bacteria ( such as Vancomycin-resistant Enterococcus，third-generation cephalosporin resistance E. coli, Methicillin-resistant Staphylococcus aureous, Extended-spectrum beta lactamase E. coli and K. pneumoniae)
  3. Changes of the bacteria virulence factors for the intestinal E. coli and K. pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Cheng Wang, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan